CLINICAL TRIAL: NCT00005537
Title: Genetics of Airway Responsiveness and Lung Function
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 5071; R01HL056371 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-08

CONDITIONS: Asthma; Lung Diseases, Obstructive; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Lung Diseases, Obstructive; Pulmonary Disease, Chronic Obstructive

SUMMARY:
To perform a genome-wide search for genes affecting two phenotypes related to asthma and chronic obstructive pulmonary disease (COPD) in a Chinese population.

DETAILED DESCRIPTION:
DESIGN NARRATIVE:

Airway responsiveness and lung function, endpoints with a strong genetic basis, are central to the obstructive airway diseases (asthma and COPD). In contrast, the dissection of the underlying genes requires unique sample resources, accurate and comprehensive phenotyping, and an efficient study design. To address to this three-pronged challenge, a genomic screen brought together a large, homogenous, mostly untreated sample from Anhui, China, a wealth of expertise in asthma phenotypes, and a potent study design based on extreme discordant sib pairs.

Since this approach utilized an extant asthmatic family population, no support for data collection was required. The primary focus of the study was two intermediate phenotypes related to asthma and COPD: airway responsiveness (characterized by increased responsiveness to histamine methacholine or other nonspecific agonists and measured by the slope of the dose response relationship) and forced expiratory volume in 1 second (FEV1). Since both traits are continuous, the appropriate study design considered only siblings with extremely discordant phenotypes. For many studies, this strategy was not feasible due to the thousands of families that must be phenotyped to identify a sample of such siblings. The plan was to utilize the organization of a well-established network in China to collect 150 extreme discordant sib pairs of each intermediate phenotype. For airway responsiveness, the estimated power from this sample, equivalent to roughly 600 concordant sib pairs, was intended to surpass the power of all existing studies, including the U.S. Collaborative Study on the Genetics of Asthma. Further, with similar power, this was the first study to test for linkage to FEV1. Moreover, to further augment power, potential phenotypic heterogeneity was reduced by stratifying the analyses by total and specific serum IgE levels, skin test reactivity, peripheral blood eosinophilia, respiratory symptoms, age, gender, bronchodilator response, and cigarette smoking.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1997-07; Study Completion 2002-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Xiping Xu — Brigham and Women's Hospital

REFERENCES:
- [Background] Hu FB, Wang B, Chen C, Jin Y, Yang J, Stampfer MJ, Xu X. Body mass index and cardiovascular risk factors in a rural Chinese population. Am J Epidemiol. 2000 Jan 1;151(1):88-97. doi: 10.1093/oxfordjournals.aje.a010127. PMID 10625178
- [Background] Xu X, Yang J, Chen C, Wang B, Jin Y, Fang Z, Wang X, Weiss ST. Familial aggregation of pulmonary function in a rural Chinese community. Am J Respir Crit Care Med. 1999 Dec;160(6):1928-33. doi: 10.1164/ajrccm.160.6.9902013. PMID 10588608
- [Background] Wang X, Wang B, Chen C, Yang J, Fang Z, Zuckerman B, Xu X. Familial aggregation of blood pressure in a rural Chinese community. Am J Epidemiol. 1999 Mar 1;149(5):412-20. doi: 10.1093/oxfordjournals.aje.a009828. PMID 10067900
- [Background] Xu X, Niu T, Chen C, Wang B, Jin Y, Yang J, Weiss ST. Association of airway responsiveness with asthma and persistent wheeze in a Chinese population. Chest. 2001 Mar;119(3):691-700. doi: 10.1378/chest.119.3.691. PMID 11243944
- [Background] Betensky RA, Hudson JI, Jones CA, Hu F, Wang B, Chen C, Xu X. A computationally simple test of homogeneity of odds ratios for twin data. Genet Epidemiol. 2001 Feb;20(2):228-38. doi: 10.1002/1098-2272(200102)20:23.0.CO;2-4. PMID 11180448
- [Background] Niu T, Rogus JJ, Chen C, Wang B, Yang J, Fang Z, Weiss ST, Xu X. Familial aggregation of bronchodilator response: a community-based study. Am J Respir Crit Care Med. 2000 Nov;162(5):1833-7. doi: 10.1164/ajrccm.162.5.9908127. PMID 11069822
- [Background] Xu X, Fang Z, Wang B, Chen C, Guang W, Jin Y, Yang J, Lewitzky S, Aelony A, Parker A, Meyer J, Weiss ST, Xu X. A genomewide search for quantitative-trait loci underlying asthma. Am J Hum Genet. 2001 Dec;69(6):1271-7. doi: 10.1086/324650. Epub 2001 Oct 22. PMID 11673820
- [Background] Venners SA, Wang X, Chen C, Wang B, Ni J, Jin Y, Yang J, Fang Z, Weiss ST, Xu X. Exposure-response relationship between paternal smoking and children's pulmonary function. Am J Respir Crit Care Med. 2001 Sep 15;164(6):973-6. doi: 10.1164/ajrccm.164.6.2009063. PMID 11587981
- [Background] Wang Z, Chen C, Niu T, Wu D, Yang J, Wang B, Fang Z, Yandava CN, Drazen JM, Weiss ST, Xu X. Association of asthma with beta(2)-adrenergic receptor gene polymorphism and cigarette smoking. Am J Respir Crit Care Med. 2001 May;163(6):1404-9. doi: 10.1164/ajrccm.163.6.2001101. PMID 11371409